CLINICAL TRIAL: NCT02860767
Title: Dosing of Antibiotics (Serum and Periprosthetic Tissues) During Reimplantation of Infected Knee and Hip Prostheses
Brief Title: Dosing of Antibiotics During Reimplantation of Infected Knee and Hip Prostheses
Acronym: DOSOS
Status: Completed | Type: Observational
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-000889-11
Record Dates: First submitted 2016-08-05; First posted 2016-08-09 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2016-08

CONDITIONS: Prosthesis-Related Infections
Keywords: Prosthesis-Related Infections; Antibiotic dosing; Reimplantation; Knee-prothesis; Hip-prothesis
MeSH Terms: conditions — Prosthesis-Related Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to evaluate the concentrations of antibiotics used as empirical treatment in serum and periprosthetic tissues during reimplantation of infected hip and knee prostheses

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the concentrations of antibiotics (daptomycin, vancomycin, cefotaxime, ceftriaxone, cefepime) in serum and periprosthetic tissues(bone and synovial joint) used as empirical treatment during reimplantation of infected hip and knee prostheses (1-stage or 2-stage management).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged of 18 years or more) who undergo reimplantation surgery for infected hip or knee prosthesis (performed in 1 or 2-stage(s)), and for whom referral physicians plans to use an empirical antibiotic therapy including cefotaxime, ceftriaxone, cefepime, daptomycin, or vancomycin.

Exclusion Criteria:

* Patients with multiple prosthetic joint infections, or with curative antibiotic therapy ongoing within two weeks or less prior to surgery, or for whom an antibiotic prophylaxis is decided by referral for the reimplantation surgery, or for whom an antibiotic-loaded cement containing the same antibiotic chosen for empirical therapy after reimplantation was used in case of 2-stage exchange

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with hip and knee prostheses infections
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-08; Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure was the evaluation of concentrations in serum and periprosthetic tissues of antibiotic agents used as empirical therapy during reimplantation of the infected prosthesis | 1 day

SECONDARY OUTCOMES:
Secondary outcome will analyze the ratio of antibiotic concentration in serum and prosthetic tissues to minimum inhibitory concentration of the concerned antibiotic for the pathogen(s) identified in intraoperative samples | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Senneville, MD, PhD, Study Director — Dron Hospital Tourcoing France; Sophie Nguyen, MD, Principal Investigator — Dron Hospital Tourcoing France
Locations (5):
- France (5):
  - CHU, Amiens
  - CHU, Caen
  - CHRU, Lille
  - CHU, Rouen
  - Dron Hospital, Tourcoing

IPD SHARING:
Plan to Share IPD: No